CLINICAL TRIAL: NCT02476110
Title: Oral Nutritive Supplements : Indications, Prescription and Follow-up for Hospitalized and Out-patients at Nutritional Risk or With Malnutrition. A Quality Care Programme at the Geneva University Hospital : The ONSHUG Survey
Brief Title: The ONSHUG Survey : A Quality Care Programme
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Professor of Nutrition and Head of Clinical Nutrition Unit, University Hospital, Geneva
Other Study IDs: Quality program ONSHUG 2015-04
Record Dates: First submitted 2015-06-01; First posted 2015-06-19 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Undernutrition
Keywords: Oral nutritive supplements; Nutritional risk screening; Homecare
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Oral nutritive supplements

SUMMARY:
Hypothesis : At hospital discharge for home, the medical prescription of ONS according to the official criteria of SSNC and the legal regulations (completed prescription according to health's insurance and homecare delivery) dictates the compliance of the patient and the reimbursement of the ONS.

DETAILED DESCRIPTION:
Rationale : At hospital admission, patients with an acute or chronically impaired nutritional balance are at nutritional risk. These patients can be identified by the Nutritional Risk Score 2002 (NRS 2002). Oral Nutritive Supplements (ONS) represent the first line of nutrition intervention. ONS are frequently prescribed during the hospital stay, and should be continued or discontinued after the hospital discharge. This latter decision should be based on officials criteria, defined by the Swiss Society for Clinical Nutrition (SSNC). To allow ONS reimbursement according to the legal regulations, all required administrative actions should be completed at the time of ONS prescription until the end of the treatment.

Center : Geneva University Hospital (HUG), site of Cluse-Roseraie.

Design : Quality control prospective observational survey.

Population : Hospitalized adults patients with Oral Nutritive Supplements (ONS). Four hundred patients to be included.

Duration : Inclusion from April to December 2015 (9 months).

Hypothesis : At hospital discharge for home, the medical prescription of ONS according to the official criteria of SSNC and the legal regulations (completed prescription according to health's insurance and homecare delivery) dictates the compliance of the patient and the reimbursement of the ONS.

Aims : The primary aim is to document the existence of an ONS medical prescription during the hospitalization and at hospital discharge for home.

The secondary aims are to describe :

* NRS 2002 score when prescribing ONS during the hospitalization, at hospital discharge for home and one month after hospital discharge for home
* Indications for ONS prescription at hospital discharge for home according to the official criteria of SSNC
* Type of ONS prescription at hospital discharge for home
* Number of ONS consumed one month after hospital discharge compared to prescription at hospital discharge
* Timing of the discontinuation of the ONS treatment
* Reasons for stopping the ONS intake.

Methods : Included are all hospitalized adults patients with ONS prescription at the HUG. Excluded are patients with ONS delivery by a homecare before the admission at the HUG or patients refusing to consume ONS or patients with major disorders of consciousness (ex : dementia) or patients unable to consume ONS (ex : dysphagia, dysfunction of upper limbs, etc.) or patients refusing to participate to the survey.

At inclusion, the comorbidities will be assessed by the Charlson Comorbidity Index. ONS prescription and nutritional risk by the NRS 2002 score will be described at hospital and at hospital discharge for home. One month after hospital discharge for home, patient's compliance to ONS will be assessed as nutritional risk by the NRS 2002 score.

Statistics : Data will be presented as mean ± standard deviation or as numbers and percentages according to the relevance, and analyzed using Chi-squared test or unpaired t-test as required.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hospitalization in medical and surgical wards of the Geneva University Hospital, site of Cluse-Roseraie
* Oral nutritive supplements prescription during hospitalization

Exclusion Criteria:

* Oral nutritive supplements delivery by a homecare before the admission in Geneva University Hospital wards, site of Cluse-Roseraie
* Patient refusal to consume oral nutritive supplements
* Major disorders of consciousness (ex : dementia)
* Physical impossibility to consume Oral nutritive supplements (ex : dysphagia, dysfunction of upper limbs, etc.)
* Patient refusal to participate to the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults patients with Oral Nutritive Supplements in medical and surgical wards of the Geneva University Hospital, site of Cluse-Roseraie
Sampling Method: Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Oral Nutritive Supplements medical prescription | Change between prescription at hospital and prescription at hospital discharge (an expected average of 6 days after admission)

SECONDARY OUTCOMES:
NRS 2002 score assessed by questionnaire | Change between score at oral nutritive supplements prescription at hospital and score at hospital discharge for home (an expected average of 6 days after admission) and score one month after hospital discharge for home
Indications for oral nutritive supplements prescription according to the official criteria of SSNC | At hospital discharge for home (an expected average of 6 days after admission)
Number of oral nutritive supplements consumed compared to prescription at hospital discharge | One month after hospital discharge
Timing for stopping the oral nutritive supplements intake if stopped | One month after hospital discharge
Reasons for stopping the oral nutritive supplements intake if stopped | One month after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Mareschal J, Altwegg J, Berthet D, Chikhi M, Chopard P, Graf S, Sierro C, Pichard C, Genton L. Prescription and indication for oral nutritional supplements in a Swiss university hospital: a prospective survey. Swiss Med Wkly. 2017 Aug 3;147:w14475. doi: 10.4414/smw.2017.14475. eCollection 2017. PMID 28804864